CLINICAL TRIAL: NCT00659776
Title: Multi-Disciplinary Study: Magnetic Resonance, Histologic And Electron Microscopy Imaging Of Intravenous Superparamagnetic Crystalline Particles (Ferumoxytol) In CNS Inflammation
Brief Title: MR, Histologic And EM Imaging Of Intravenous Ferumoxytol In Central Nervous System (CNS) Inflammation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to staffing shortages and lack of funding during Covid.
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OHSU-1562; 5R01NS034608 (NIH)
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Nervous System Diseases; Diagnostic Imaging
Keywords: ferumoxytol
MeSH Terms: conditions — Nervous System Diseases | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Inflammatory lesions (Active Comparator): Subjects with dural, central nervous system (CNS) parenchymal based inflammatory, vascular or demyelinating lesions.
  Interventions: Drug: Ferumoxytol
- Vascular lesions (Active Comparator): subjects will include those with vascular CNS lesions such as ischemic stroke, transient ischemic attack (TIA) with suspected carotid embolic origin, or vasculopathy involving the carotids, (including diagnosed carotid stenosis >50%) the aorta, or the arteries of the extremities, or diagnosed thrombosis of the intraabdominal, pelvic or extremity veins.
  Interventions: Drug: Ferumoxytol
- Lymph nodes (Active Comparator): Subjects with enlarged cervical lymph nodes in which inflammatory processes (reactive lymph nodes) is part of the differentials.
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — Ferumoxytol will be injected as i.v. bolus(es) at 3ml/s followed by a saline flush. The maximum total dose over 30 to 60 minutes will be 510mg Fe. Separate boluses will be used for perfusion MR and MRA. Ferumoxytol may be diluted up to 28 fold in normal saline to reduce T2* effects in the MR angiography. Rate of administration can be varied based on the subject's iv site, but will never exceed 510mg Fe /17s (as was done in phaseIII trials)
  Other Names: Feraheme

SUMMARY:
This exploratory study utilizes ferumoxytol, an iron oxide nanoparticle MR contrast agent for imaging various inflammatory processes in the head and neck region, spine, including the central nervous system. The protocol enrolls subjects with radiological or histological diagnosis of unknown, dural, or parenchymal CNS lesions, multiple sclerosis, TIA or stroke, vasculitis, or other vascular lesions; arterial vasculopathy and venous thrombosis; or enlarged cervical lymph nodes. The main purpose of this study is to better understand the underlying cellular mechanisms, contrast agent extravasation, uptake into macrophages and to assess its value in clinical MR imaging.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinical, radiological or established histological diagnosis of dural or central nervous system (CNS) parenchymal based inflammatory, vascular or demyelinating lesions, radiological suspected diagnosis of vascular CNS lesions such as ischemic stroke, TIA with suspected carotid embolic origin, or vasculopathy involving the carotids (including diagnosed carotid stenosis >50%), the aorta, the arteries of the extremities, or diagnosed thrombosis of the intraabdominal, pelvic or extremity veins, or clinical or radiological diagnosis of enlarged cervical lymph nodes in which inflammatory processes (reactive lymph nodes) is part of the differentials.
* Subjects must be 18 years or older
* Subjects will be followed for at least 1 month after the infusion of ferumoxytol.
* All subjects or their authorized representative must sign a written informed consent and give HIPAA authorization in accordance with institutional guidelines.
* Female subjects of child-bearing potential must be postmenopausal, surgically sterile, or using a reliable form of contraception for at least a month. These criteria can be waved at the discretion of the investigator if the one-month wait required is not in the best interest of the patient.
* Karnofsky must be 30% or greater

Exclusion Criteria:

* Subjects with clinically significant signs of uncal herniation
* Subjects who have a contraindication for MRI: metal in their bodies (a cardiac pacemaker or other incompatible device), are severely agitated, or have an allergy to Gd contrast material.
* Subjects with known allergic or hypersensitivity reactions to parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations
* Subjects with known hepatic insufficiency or cirrhosis
* Subjects with known or suspected iron overload
* HIV-positive subjects on combination anti-retroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ferumoxytol
* Pregnant or lactating women are excluded from this study because of possible risk to the fetus or infant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Inflammatory Lesions: Subjects with dural, central nervous system (CNS) parenchymal based inflammatory, vascular or demyelinating lesions.
- Group 2: Vascular Lesions: Subjects with vascular lesions
- Group 3: Lymph Nodes: Subjects with enlarged cervical lymph nodes in which inflammatory processes (reactive lymph nodes) is part of the differentials.
Period: Overall Study
Arm/Group | Group 1: Inflammatory Lesions | Group 2: Vascular Lesions | Group 3: Lymph Nodes
Started | 230 | 25 | 0
Number of Lesions Gadolinium | 145 | 0 | 0
Number of Lesions Ferumoxytol | 152 | 0 | 0
Degree of Contrast Enhancement Gadolinium | 128 | 0 | 0
Degree of Contrast Enhancement Ferumoxytol | 131 | 0 | 0
Border Delineation Gadolinium | 128 | 0 | 0
Border Delineation Ferumoxytol | 131 | 0 | 0
Internal Morphology of Lesions Gadolinium | 128 | 0 | 0
Internal Morphology of Lesions Ferumoxytol | 131 | 0 | 0
Completed | 218 | 23 | 0
Not Completed | 12 | 2 | 0
Not completed — Withdrawal by Subject | 12 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated early due to Covid and funding shortages. Therefore, subject enrollment was not met, and no subjects were enrolled in group 3.
Groups:
- Group 2: Vascular Lesions: Subjects will include those with vascular CNS lesions such as ischemic stroke, TIA with suspected carotid embolic origin, or atherosclerotic or inflammatory vasculopathy involving the carotids (including diagnosed carotid stenosis >50%), aorta and the arteries of the extremities or thrombosis of the intraabdominal, pelvic or extremity veins.
- Total: Total of all reporting groups
Arm/Group | Group 1: Inflammatory Lesions | Group 2: Vascular Lesions | Group 3: Lymph Nodes | Total
Number analyzed (Participants) | 230 | 25 | 0 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 184 | 24 |  | 208
  >=65 years | 46 | 1 |  | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (15.8) | 61.4 (9.6) |  | 52.3 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 14 |  | 119
  Male | 125 | 11 |  | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 1 |  | 17
  Not Hispanic or Latino | 213 | 24 |  | 237
  Unknown or Not Reported | 1 | 0 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 |  | 2
  Asian | 6 | 0 |  | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 3 | 0 |  | 3
  White | 213 | 25 |  | 238
  More than one race | 4 | 0 |  | 4
  Unknown or Not Reported | 2 | 0 |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 230 | 25 |  | 255

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions
Time Frame: 72 hours
Population: Due to the study closing prematurely, the images for the 23 subjects in group 2 were collected but not processed for analysis, and no data were collected in group 3 for this measure.
Measure: Mean (Standard Deviation); unit: Number of lesions
Arm/Group | Group 1: Inflammatory Lesions | Group 2: Vascular Lesions | Group 3: Lymph Nodes
Number analyzed (Participants) | 152 | 0 | 0
Number of lesions
  Gadolinium: number analyzed (Participants) | 145 | 0 | 0
  Gadolinium | 1.8 (1.17) |  |
  Ferumoxytol | 1.9 (1.09) |  |

2. Primary Outcome: Degree of Contrast Enhancement
Description: Scoring system for parameters: Degree of contrast enhancement (1=none, 2=moderate, 3=good, 4=excellent)
Time Frame: 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score of contrast enhancement
Arm/Group | Group 1: Inflammatory Lesions | Group 2: Vascular Lesions | Group 3: Lymph Nodes
Number analyzed (Participants) | 131 | 0 | 0
Score of contrast enhancement
  Gadolinium: number analyzed (Participants) | 128 | 0 | 0
  Gadolinium | 2.9 (1.13) |  |
  Ferumoxytol | 2.7 (1.13) |  |

3. Primary Outcome: Assessment of Border Delineation
Description: The scoring parameters were: (1=none, 2=moderate, 3=good, 4=excellent).
Time Frame: 72hrs
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score assessment of border delineation
Arm/Group | Group 1: Inflammatory Lesions | Group 2: Vascular Lesions | Group 3: Lymph Nodes
Number analyzed (Participants) | 131 | 0 | 0
Score assessment of border delineation
  Gadolinium: number analyzed (Participants) | 128 | 0 | 0
  Gadolinium | 3.2 (.87) |  |
  Ferumoxtyol | 3.2 (.75) |  |

4. Primary Outcome: Internal Morphology of Lesions
Description: The scoring parameters were: (1=poor, 2=moderate, 3=good).
Time Frame: 72hrs
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score of internal morphology of lesions
Units Other Than Participants: Lesion
Arm/Group | Group 1: Inflammatory Lesions | Group 2: Vascular Lesions | Group 3: Lymph Nodes
Number analyzed (Participants) | 131 | 0 | 0
Number analyzed (Lesion) | 131 | 0 | 0
Score of internal morphology of lesions
  Gadolinium: number analyzed (Participants) | 128 | 0 | 0
  Gadolinium | 2.4 (1.04) |  |
  Ferumoxytol | 2.5 (.99) |  |

5. Secondary Outcome: Ferumoxytol Particles With Histology and Electron Microscopy in Biopsy Samples
Time Frame: 72 hours
Population: Due to the study closing prematurely, we did not collect these data.
Arm/Group | Group 1: Inflammatory Lesions | Group 2: Vascular Lesions | Group 3: Lymph Nodes
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Side Effects/Safety of Ferumoxytol When Given During MRI.
Description: Number of serious adverse events attributable to ferumoxytol.
Time Frame: 30 days
Population: Of the 230 subjects enrolled in group 1, 12 withdrew or were taken of study prior to receiving ferumoxytol. The 218 subjects remaining were analyzed. Of the 25 subjects enrolled in group 2, 2 withdrew or were taken of study prior to receiving ferumoxyotol. The 23 subjects remaining were analyzed.
Measure: Number; unit: Number of serious AEs attributable to Fe
Arm/Group | Group 1: Inflammatory Lesions | Group 2: Vascular Lesions | Group 3: Lymph Nodes
Number analyzed (Participants) | 218 | 23 | 0
Number of serious AEs attributable to Fe | 1 | 0 |

7. Secondary Outcome: Iron Uptake and Clearance in Abdominal Organs, Such as the Liver, Spleen, Pancreas and Bone Marrow by Applying Usual Abdominal MR Sequences at Multiple Time Points
Time Frame: 6 months
Population: Due to the study closing prematurely, we did not enroll any subjects into this subgroup nor gather any data.
Arm/Group | Group 1: Inflammatory Lesions | Group 2: Vascular Lesions | Group 3: Lymph Nodes
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From time of ferumoxytol infusion through 30 days after ferumoxytol infusion.
Description: The SAEs reported here are all AEs of grades 3, and 4. The study was terminated early due to Covid and funding shortages. Therefore, subject enrollment was not met, and no subjects were enrolled in group 3.
Groups:
- Group 1: Inflammatory Lesions: Subjects with dural, central nervous system (CNS) parenchymal based inflammatory, vascular or demyelinating lesions.
  Ferumoxytol: Ferumoxytol will be injected as i.v. bolus(es) at 3ml/s followed by a saline flush. The maximum total dose over 30 to 60 minutes will be 510mg Fe. Separate boluses will be used for perfusion MR and MRA. Ferumoxytol may be diluted up to 28 fold in normal saline to reduce T2* effects in the MR angiography. Rate of administration can be varied based on the subject's iv site, but will never exceed 510mg Fe /17s (as was done in phaseIII trials)
- Group 2: Vascular Lesions: Subjects with vascular lesions
  Ferumoxytol: Ferumoxytol will be injected as i.v. bolus(es) at 3ml/s followed by a saline flush. The maximum total dose over 30 to 60 minutes will be 510mg Fe. Separate boluses will be used for perfusion MR and MRA. Ferumoxytol may be diluted up to 28 fold in normal saline to reduce T2* effects in the MR angiography. Rate of administration can be varied based on the subject's iv site, but will never exceed 510mg Fe /17s (as was done in phaseIII trials)
- Group 3: Lymph Nodes: Subjects with enlarged cervical lymph nodes in which inflammatory processes (reactive lymph nodes) is part of the differentials.
  Ferumoxytol: Ferumoxytol will be injected as i.v. bolus(es) at 3ml/s followed by a saline flush. The maximum total dose over 30 to 60 minutes will be 510mg Fe. Separate boluses will be used for perfusion MR and MRA. Ferumoxytol may be diluted up to 28 fold in normal saline to reduce T2* effects in the MR angiography. Rate of administration can be varied based on the subject's iv site, but will never exceed 510mg Fe /17s (as was done in phaseIII trials)
Arm/Group | Group 1: Inflammatory Lesions | Group 2: Vascular Lesions | Group 3: Lymph Nodes
All-Cause Mortality (participants affected / at risk) | 1/218 | 0/23 | 0/0
Serious Adverse Events (participants affected / at risk) | 39/218 | 2/23 | 0/0
Other Adverse Events (participants affected / at risk) | 11/218 | 2/23 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Inflammatory Lesions (N=218) | Group 2: Vascular Lesions (N=23) | Group 3: Lymph Nodes (N=0)
Ataxia (Nervous system disorders) | 8 (8) | 0 (0) | 0 (0)
Back Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage (Investigations) | 1 (1) | 0 (0) | 0 (0) — CNS hemorrhage
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
DVT (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever with ANC<1 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 6 (6) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0)
Pulmonary embolus (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Speech impairment (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Pain at surgical site (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Inflammatory Lesions (N=218) | Group 2: Vascular Lesions (N=23) | Group 3: Lymph Nodes (N=0)
Nausea (Gastrointestinal disorders) | 11 (11) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT00659776/Prot_SAP_000.pdf